CLINICAL TRIAL: NCT07030348
Title: Early Diagnosis of Pancreatic Cancer Duodenal Fluid-Based Biomarker Exploratory Study
Status: Recruiting | Type: Observational
Sponsor: Do Hyun Park (Other)
Collaborators: The Cleveland Clinic (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor-Investigator, Do Hyun Park, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: DHP_Bio; AMC_IRB_2023-1498 (Other: Asan Medical Center Institutional Review Board)
Record Dates: First submitted 2025-05-21; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancers; Pancreatic Diseases
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 263
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic Cancer Group (DP): Participants with a biopsy with proven stage I-IV pancreatic ductal adenocarcinoma (PDAC), or with suspected pancreatic cancer on imaging and scheduled for an endoscopic ultrasound-guided pancreatic biopsy.
- Non-Pancreatic Cancer Group (DC): Participants with pancreatic cystic tumors or with acute or chronic pancreatitis, or with no evidence of a pancreatic disease

SUMMARY:
Purpose Pancreatic cancer is the fourth leading cancer-related mortality disease in the United States, with a five-year survival rate of 11%, and only 10 15% of all pancreatic cancer patients are operable or borderline operable.

Therefore, there is an unmet need for early diagnosis of pancreatic cancer; however, biomarkers related to this are not well understood. This study aims to identify biomarkers for the early diagnosis of pancreatic cancer through duodenal pancreatic juice, which can be easily obtained through an endoscopy.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cancer-related mortality disease in the United States, with a five-year survival rate of 11%, which is a very poor prognosis, and only 10-15% of all pancreatic cancer patients are operable or borderline operable.

Therefore, there is an unmet need for early diagnosis of pancreatic cancer; however, the biomarkers of humoral fluids associated with the early diagnosis of pancreatic cancer are not well understood.

Duodenal pancreatic fluids can be easily obtained through an endoscopy and contain a large amount of pancreatic fluid secreted by the pancreas, which is known to be a candidate of biomarkers for early diagnosis of pancreatic cancer.

However, there have been few studies using duodenal fluids in Korea. This study aims to prospectively analyze biomarkers for early diagnosis of pancreatic cancer using duodenal fluids obtained by endoscopy in pancreatic and non-pancreatic cancer groups.

ELIGIBILITY:
Inclusion Criteria:

Among the patients requiring gastro-duodenal endoscopy, endoscopic ultrasound, or ERCP for medical purposes, the pancreatic cancer group should meet the criteria numbered 1, 2, and either 3 or 4.

1. Be at least 19 years old.
2. Have completed the informed consent for planned upper endoscopy, endoscopic ultrasound, or endoscopic retrograde cholangiopancreatography before the duodenal fluid collection.
3. A biopsy with proven stage I-IV pancreatic ductal adenocarcinoma (PDAC).
4. Suspected pancreatic cancer on imaging and scheduled for an endoscopic ultrasound-guided pancreatic biopsy.

The non-pancreatic cancer group should meet the criteria numbered 1, 2, and either 3 or 4.

1. Be at least 19 years old.
2. Have completed the informed consent for planned upper endoscopy, endoscopic ultrasound, or endoscopic retrograde cholangiopancreatography before the duodenal fluid collection.
3. Patients with pancreatic cystic tumors or patients with acute or chronic pancreatitis.
4. No evidence of a pancreatic disease.

Exclusion Criteria:

The exclusion criteria for the pancreatic cancer and the non-pancreatic cancer groups will be:

1. Innate or post-surgical anatomy that precludes direct sampling of duodenal fluid.
2. Hemodynamically unstable and unable to have an endoscopy performed.
3. A large amount of ascites fluid that is not controlled and unable to have an endoscopy performed.
4. A coagulation disorder that cannot be corrected and unable to have an endoscopy performed.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who require a gastro-duodenal endoscopy, endoscopic ultrasound, or endoscopic retrograde cholangiopancreatography (ERCP) for medical purposes will be enrolled in this study. The pancreatic cancer group and the control non-pancreatic cancer group will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of Biomarkers for Early Pancreatic Cancer Detection | Up to 1 year from baseline
  Area Under the Receiver Operating Characteristic Curve (AUC) and 95% Confidence Interval (CI) of candidate biomarkers in the training cohort. If the AUC falls within ±5% of the target value (0.94), the optimal cutoff value for pancreatic cancer differentiation will be reported using Youden's Index.

SECONDARY OUTCOMES:
External Validation Using U.S. Samples | Up to 2 year from baseline
  Area under the ROC curve (AUC) of candidate biomarkers in the U.S. validation cohort using cut-off values derived from the Korean training cohort

OTHER OUTCOMES:
Optimizing Sample Collection Volume | Up to 6 month from baseline
  Correlation between duodenal fluid sample volume (mL) and biomarker detection sensitivity (AUC or concentration)
Assessing Racial Differences in Biomarker Expression | Up to 2 year from baseline
  Mean biomarker expression levels in Korean vs. U.S. cohorts as measured in duodenal fluid samples
Evaluating the Impact of Secretin Administration | Up to 1 year from baseline
  Comparison of biomarker concentrations in duodenal fluid with vs. without secretin stimulation
Longitudinal Analysis of non-pancreatic cancer group Samples (Asan Medical Center Only) | Up to 2 year from baseline
  Change in biomarker levels between first and second duodenal fluid samples in non-pancreatic cancer participants

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Cleveland Clinic, Cleveland, Ohio
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No